CLINICAL TRIAL: NCT00759330
Title: A Multi-Center, Randomized, Double-Blind, Placebo-Controlled Trial of Flurbiprofen Tape for Treatment of Chronic Low Back Pain
Brief Title: Flurbiprofen Tape for Treatment of Chronic Low Back Pain
Acronym: LBP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teikoku Pharma USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TPU FT-US06-01; NCT00759330 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Results first posted 2016-10-06 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-06

CONDITIONS: Chronic Low Back Pain
Keywords: Flurbiprofen, low back pain, chronic low back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo Tape (Arm 1) (Placebo Comparator): Placebo tape remained on for 12 hours of continuous treatment per day.
  Interventions: Drug: Placebo Tape (Arm 1)
- Flurbiprofen Tape (Arm 2) (Experimental): Flurbiprofen tape remained on for 12 hours of continuous treatment per day.
  Interventions: Drug: Flurbiprofen Tape (Arm 2)
- Placebo Tape (Arm 3) (Placebo Comparator): Placebo tape remained on for 24 hours of continuous treatment per day.
  Interventions: Drug: Placebo Tape (Arm 3)
- Flurbiprofen Tape (Arm 4) (Experimental): Flurbiprofen tape remained on for 24 hours of continuous treatment per day.
  Interventions: Drug: Flurbiprofen Tape (Arm 4)

INTERVENTIONS:
Drug: Placebo Tape (Arm 1) — Two placebo tapes (one on each side of the spine) were applied on the lower back area once daily for 7 days.
  Arms: Placebo Tape (Arm 1)
Drug: Flurbiprofen Tape (Arm 2) — Two flurbiprofen tapes (one on each side of the spine) were applied on the lower back area once daily for 7 days. Each tape contained 31.5 mg flurbiprofen for a total daily dose of 63 mg.
  Arms: Flurbiprofen Tape (Arm 2)
Drug: Placebo Tape (Arm 3) — Two placebo tapes (one on each side of the spine) were applied on the lower back area once daily for 7 days.
  Arms: Placebo Tape (Arm 3)
Drug: Flurbiprofen Tape (Arm 4) — Two flurbiprofen tapes (one on each side of the spine) were applied on the lower back area once daily for 7 days. Each tape contained 31.5 mg flurbiprofen for a total daily dose of 63 mg.
  Arms: Flurbiprofen Tape (Arm 4)

SUMMARY:
The purpose of this trial is to evaluate the analgesic efficacy and safety of flurbiprofen tape for chronic low back pain (lasting greater than 3 months).

DETAILED DESCRIPTION:
This study is a multi-center, randomized, double-blind, placebo-controlled study in patients with daily low back pain below the 12th thoracic vertebra of greater than 3 months duration. Patients also had an average daily pain score of 4 or greater on an 11-point categorical pain scale for the last 3 days of the baseline phase. The study began with a 14-day washout period of previously used pain medications. At the end of the 14-day baseline phase, patients were randomized to 1 of 4 treatments: Flurbiprofen tape applied once daily for 12 hours, Flurbiprofen tape applied once daily for 24 hours, placebo tape applied once daily for 12 hours, or placebo tape applied once daily for 24 hours. During the 7-day treatment phase, patients applied 2 treatment tapes once daily for 7 days. The tapes remained on for 12 or 24 hours of continuous treatment, depending on the treatment to which they were randomized. Patients were provided with rescue medication. After 7 days of tape treatment, patients returned to the clinic for a study exit visit.

ELIGIBILITY:
Inclusion Criteria:

* male or female 18 to 80 years;
* signed an informed consent;
* daily LBP below the 12th thoracic vertebra of greater than 3 months' duration;
* able to ambulate at least 100 meters;
* in stable general health with laboratory values within normal limits
* no evidence of drug abuse or residual opiates; determined by urine drug screening;
* diagnosis of chronic LBP verified by medical records;
* female patients must be postmenopausal (defined as 1 year without menses), physically incapable of becoming pregnant, or using an acceptable birth control method. Non-postmenopausal patients must have confirmation of a negative urine pregnancy test;
* must read and speak English;
* must be reliable and mentally competent to complete study measurements;
* must be available for the study visits and telephone checks from study entry to study completion.
* male patients must use an acceptable method of birth control with their female partners;
* rates their pain at 3 or higher on an 11-point Categorical Pain Scale for LBP over the prior week (7 days) of Visit 1.
* over the last 3 days of the Baseline Phase, had a computed average pain score of 4 or greater on an 11-point Categorical Pain Scale
* discontinued the use of any topical pain medications, salves, anticonvulsants, oral NSAIDs, muscle relaxants, opioids, or anti-inflammatory steroids during the Baseline Phase. Acetaminophen, at a dose of ≤ 1000 mg per day is acceptable;
* able to discontinue the use of therapy defined as ice, heat, chiropractic care, physical therapy, acupuncture and acupressure on their lower back area during the Baseline Phase.

Exclusion Criteria:

* open skin lesion within the painful area;
* experiencing LBP for less than 3 months;
* undergone back surgery within the past 3 months or has plans for back surgery within 30 days post-study;
* participated in clinical treatment studies within 30 days of study entry;
* chronic back pain which is due to fibromyalgia or connective tissue disorder (lupus, rheumatoid arthritis, ankylosing spondylitis, Reiter's syndrome, etc.);
* LBP due to malignancy, vertebral fracture, or infection;
* used opioids (including low potency/low dose opioid combinations and tramadol) more than 2 times per week within 30 days of study entry. Opioids and tramadol must not have been taken at least 4 days prior to study entry;
* had injection therapy within 30 days of study entry, including corticosteroids;
* a clinically significant psychiatric disorder (severe depression, other Axis I or Axis II disorders as defined in the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV);
* taking lithium, furosemide, and/or thiazides;
* considered unreliable as to medication compliance (if any medication other than 1000 mg or less of acetaminophen a day was taken for any type of pain, the patient was discontinued) or adherence to scheduled appointments as determined by the investigators;
* a prior history of GI bleeds/ulcers or clinically significant liver/kidney disease;
* known hypersensitivity to flurbiprofen or other NSAIDs;
* has a coagulation disorder or is taking warfarin or other anticoagulants (aspirin at a dose of [≤ 81 mg] is acceptable);
* clinically significant fluid retention, cardiovascular disease (CVD), hypertension, or heart failure;
* had coronary artery bypass graft surgery (CABG), cardiovascular thrombotic event, myocardial infarction (MI) and/or stroke within 1 year of Visit 1;
* had unresolved litigation related to back injury or other pain complaints; settled disability claims/payments (Worker's Compensation, state/federal/private disability plans) were allowed.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2007-10; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Song, Study Director — Teikoku Pharma USA, Inc.
Locations (10):
- United States (10):
  - Redpoint Research, Phoenix, Arizona
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - University Foundation for Education and Research, Inc., Tampa, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Internal Medicine Associates of Cordova, Cordova, Tennessee
  - Sarah Cannon Research Institute, Memphis, Tennessee
  - Senior Adults Specialty Research, Austin, Texas
  - Charolettesville Medical Research, Charlottesville, Virginia
  - Rainier Clinical Research Center, Inc., Renton, Washington
  - Aurora Advanced Healthcare, Inc., Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 10 clinical sites in the US from September 2007 to July 2008. Patients with chronic LBP below the 12th thoracic vertebra of greater than 3 months duration and with an average daily pain score of 4 or greater on an 11-point categorical pain scale for the last 3 days of the baseline phase were eligible to participate.
Pre-assignment Details: Prior to randomization into the Tape Treatment Phase, participants began a 14-day washout period of previously used pain medications. Participants were then randomized to 1 of 4 treatments. After 7 days of treatment, patients returned to the clinic for a study exit visit. Participants were provided with rescue medication throughout the study.
Groups:
- Placebo Tape, Daily for 12 Hours: Two placebo tapes (one on each side of the spine) were applied on the lower back area once daily for 7 days. The tapes remained on for 12 hours of continuous treatment per day.
- Flurbiprofen Tape, Daily for 12 Hours: Two flurbiprofen tapes (one on each side of the spine) were applied on the lower back area once daily for 7 days. The tapes remained on for 12 hours of continuous treatment per day. Each tape contained 31.5 mg flurbiprofen for a total daily dose of 63 mg.
- Placebo Tape, Daily for 24 Hours: Two placebo tapes (one on each side of the spine) were applied on the lower back area once daily for 7 days. The tapes remained on for 24 hours of continuous treatment per day.
- Flurbiprofen Tape, Daily for 24 Hours: Two flurbiprofen tapes (one on each side of the spine) were applied on the lower back area once daily for 7 days. The tapes remained on for 24 hours of continuous treatment per day. Each tape included 31.5 mg flurbiprofen for a total daily dose of 63 mg.
Period: Overall Study
Arm/Group | Placebo Tape, Daily for 12 Hours | Flurbiprofen Tape, Daily for 12 Hours | Placebo Tape, Daily for 24 Hours | Flurbiprofen Tape, Daily for 24 Hours
Started | 20 | 42 | 22 | 43
Completed | 19 | 41 | 22 | 41
Not Completed | 1 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Flurbiprofen Tape, Daily for 24 Hours: Two flurbiprofen tapes (one on each side of the spine) were applied on the lower back area once daily for 7 days. The tapes remained on for 24 hours of continuous treatment per day. Each tape contained 31.5 mg flurbiprofen for a total daily dose of 63 mg.
- Total: Total of all reporting groups
Arm/Group | Placebo Tape, Daily for 12 Hours | Flurbiprofen Tape, Daily for 12 Hours | Placebo Tape, Daily for 24 Hours | Flurbiprofen Tape, Daily for 24 Hours | Total
Number analyzed (Participants) | 20 | 42 | 22 | 43 | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (14.47) | 50.1 (13.02) | 53.6 (13.46) | 53.0 (11.98) | 52.1 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 23 | 9 | 28 | 69
  Male | 11 | 19 | 13 | 15 | 58

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Summed Pain Intensity Difference (SPID+)
Description: The primary efficacy endpoint was the cumulative summed pain intensity difference (SPID+) at Days 4 and 7 of the tape treatment phase as computed from the daily categorical pain scale score reported on the patient's daily diary during the tape treatment phase; pain was rated on an 11-point scale, where: 0 = no pain, 10 = worst pain imaginable.
  Summed pain intensity difference is the sum of the pain intensity differences (PID). PID at each post-baseline evaluation was computed as the average baseline categorical pain scale score minus the post-baseline categorical pain scale score from the daily dairy. For patients with multiple pain scores reported on a given post-baseline study day, the PID scores were averaged to compute one daily PID score for each patient.
Time Frame: Days 4 and 7 of tape treatment phase
Population: Reported data are based on Intent-to-Treat patient population.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Tape, Daily for 12 Hours | Flurbiprofen Tape, Daily for 12 Hours | Placebo Tape, Daily for 24 Hours | Flurbiprofen Tape, Daily for 24 Hours
Number analyzed (Participants) | 20 | 42 | 22 | 43
units on a scale
  SPID for Day 4 | 4.6 (1.62) | 6.3 (1.14) | 6.7 (1.56) | 5.2 (1.13)
  SPID for Day 7 | 8.4 (2.95) | 12.1 (2.06) | 13.0 (2.82) | 10.2 (2.05)

2. Secondary Outcome: Pain Intensity Difference (PID+)
Description: +PID = pre-treatment value at baseline - post-treatment value at day of evaluation, where: pre-treatment value at baseline = average daily pain over the last 3 days of the baseline phase (ie, average of daily averages of the categorical pain scale scores for the last 3 days of the baseline phase). Pain was rated on an 11-point scale, where: 0 = no pain, 10 = worst pain imaginable.
  A positive PID indicates a reduction in pain.
Time Frame: Days 1 through 7 of tape treatment phase
Population: Reported data are based on Intent-to-Treat patient population.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Tape, Daily for 12 Hours | Flurbiprofen Tape, Daily for 12 Hours | Placebo Tape, Daily for 24 Hours | Flurbiprofen Tape, Daily for 24 Hours
Number analyzed (Participants) | 20 | 42 | 22 | 43
units on a scale
  Day 1 | 0.9 (0.38) | 1.3 (0.26) | 1.1 (0.36) | 0.8 (0.26)
  Day 2 | 1.4 (0.46) | 1.3 (0.32) | 1.8 (0.44) | 1.4 (0.32)
  Day 3 | 1.2 (0.48) | 1.6 (0.34) | 2.0 (0.46) | 1.6 (0.33)
  Day 4 | 1.1 (0.49) | 2.1 (0.34) | 1.8 (0.47) | 1.4 (0.34)
  Day 5 | 1.1 (0.49) | 1.7 (0.34) | 2.1 (0.47) | 1.5 (0.34)
  Day 6 | 1.2 (0.50) | 1.9 (0.35) | 2.0 (0.48) | 1.5 (0.35)
  Day 7 | 1.6 (0.52) | 2.2 (0.36) | 2.2 (0.49) | 1.9 (0.36)

3. Secondary Outcome: Average Daily Categorical Pain Scale Scores
Description: Patients rated their lower back pain, caused by normal activity and movement, on an 11-point categorical pain scale, where:
  0 = no pain, and 10 = worst pain imaginable. Patients rated their lower back pain every 12 hours, at any time they took medication including rescue medication for any type of pain, and if they applied or removed their treatment tapes at a time other than the scheduled time.
  Data are reported as the daily average categorical pain scale score by treatment group.
Time Frame: Days 1 through 7 of tape treatment phase
Population: Reported data are based on Intent-to-Treat patient population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Tape, Daily for 12 Hours | Flurbiprofen Tape, Daily for 12 Hours | Placebo Tape, Daily for 24 Hours | Flurbiprofen Tape, Daily for 24 Hours
Number analyzed (Participants) | 20 | 42 | 22 | 43
units on a scale
  Day 1 | 5.3 (2.10) | 4.8 (1.92) | 5.3 (2.18) | 5.7 (1.85)
  Day 2 | 4.7 (2.37) | 4.7 (1.96) | 4.5 (2.26) | 4.9 (2.51)
  Day 3 | 5.0 (2.65) | 4.5 (2.04) | 4.3 (2.36) | 4.8 (2.39)
  Day 4 | 5.0 (2.57) | 4.0 (2.20) | 4.5 (2.59) | 5.0 (2.54)
  Day 5 | 5.1 (2.74) | 4.4 (2.56) | 4.2 (2.38) | 4.8 (2.44)
  Day 6 | 4.9 (2.78) | 4.2 (2.46) | 4.2 (2.43) | 4.8 (2.60)
  Day 7 | 4.6 (2.55) | 3.8 (2.33) | 4.1 (2.50) | 4.4 (2.59)

4. Secondary Outcome: Percent Change From Baseline in Total Functional Rating Index (FRI)
Description: Patients completed the FRI, a 10-item back pain-specific measure of function questionnaire describing the condition at the time the questionnaire was completed; each item (pain intensity, sleeping, personal care, travel, etc.) was rated on a 5-point scale, where 0 = best outcome, 4 = worst outcome.
  FRI was reported as the percent change from baseline at Day 7 of the tape treatment phase, where:
  Total FRI score = sum of the 10 questions. The total FRI score ranged from 0 (best outcome) to 40 (worst outcome). Percent change = ([baseline - Day 7]/baseline)*100.
  A positive percent change indicates a favorable treatment effect.
Time Frame: baseline to Day 7 of tape treatment phase
Population: Reported data are based on Intent-to-Treat patient population. Discrepancy in the number of participants analyzed for this outcome measure is due to discontinuations: 1 participant in the placebo tape12 hour group and 2 participants in the flurbiprofen tape groups (1 in the 12 hour group and 1 in the 24 hour group).
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | Placebo Tape, Daily for 12 Hours | Flurbiprofen Tape, Daily for 12 Hours | Placebo Tape, Daily for 24 Hours | Flurbiprofen Tape, Daily for 24 Hours
Number analyzed (Participants) | 19 | 41 | 22 | 42
percent change from baseline | 20.6 (7.40) | 29.0 (5.10) | 28.2 (6.93) | 25.4 (5.10)

5. Secondary Outcome: Change From Baseline in Total Tender Point Examination Score
Description: At baseline and Day 7 of the tape treatment phase, patients had an assessment of tenderness bilaterally at the sacroiliac joint, greater trochanter of the hip, gluteus medius and minimus, and paraspinal muscles at L3-L4, L4-L5, and L5-S1. The investigator or research nurse pressed 12 specific areas of the body (6 locations, left and right sides), and patients were asked to rate the intensity of their pain at those 12 areas using an 11-point scale, where:
  0 = no pain, 10 = the worst pain the patient has ever experienced. The total tender point examination score ranged from 0 (best outcome) to 120 (worst outcome). Change from baseline = baseline - Day 7. A positive change indicates a favorable treatment effect.
Time Frame: Baseline to Day 7 of tape treatment phase
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo Tape, Daily for 12 Hours | Flurbiprofen Tape, Daily for 12 Hours | Placebo Tape, Daily for 24 Hours | Flurbiprofen Tape, Daily for 24 Hours
Number analyzed (Participants) | 19 | 41 | 22 | 42
units on a scale | 13.9 (4.40) | 11.7 (3.03) | 19.2 (4.12) | 9.2 (3.03)

6. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: At Day 7, patients provided their PGIC with regard to lower back pain response to treatment, using a 7-point scale, where:
  1 = very much improved, 7 = very much worse.
Time Frame: Day 7
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Placebo Tape, Daily for 12 Hours | Flurbiprofen Tape, Daily for 12 Hours | Placebo Tape, Daily for 24 Hours | Flurbiprofen Tape, Daily for 24 Hours
Number analyzed (Participants) | 19 | 41 | 22 | 42
participants
  1: Very much improved | 3 | 7 | 3 | 9
  2: Much improved | 1 | 10 | 3 | 4
  3: Improved | 4 | 12 | 8 | 11
  4: No change | 10 | 10 | 8 | 18
  5: Worse | 1 | 2 | 0 | 0
  6: Much worse | 0 | 0 | 0 | 0
  7: Very much worse | 0 | 0 | 0 | 0

7. Secondary Outcome: Acetaminophen Used During the Tape Treatment Phase
Description: The percentage of patients who used rescue medication during the tape treatment phase.
Time Frame: Day 1 through Day 7 of the tape treatment phase
Population: Reported data are based on Intent-to-Treat patient population.
Measure: Number; unit: percentage of patients
Arm/Group | Placebo Tape, Daily for 12 Hours | Flurbiprofen Tape, Daily for 12 Hours | Placebo Tape, Daily for 24 Hours | Flurbiprofen Tape, Daily for 24 Hours
Number analyzed (Participants) | 20 | 42 | 22 | 43
percentage of patients | 50 | 54.8 | 36.4 | 62.8

8. Secondary Outcome: Acetaminophen Used During the Tape Treatment Phase
Description: The total amount (mg) of rescue medication used during the tape treatment phase.
Time Frame: Day 1 through Day 7 of the tape treatment phase
Population: Reported data are based on Intent-to-Treat patient population.
Measure: Least Squares Mean (Standard Error); unit: mg
Arm/Group | Placebo Tape, Daily for 12 Hours | Flurbiprofen Tape, Daily for 12 Hours | Placebo Tape, Daily for 24 Hours | Flurbiprofen Tape, Daily for 24 Hours
Number analyzed (Participants) | 20 | 42 | 22 | 43
mg | 2226.9 (537.6) | 1617.5 (376.0) | 1585.4 (515.2) | 2141.3 (373.5)

9. Secondary Outcome: Percentage of Patients Who Discontinued
Description: The percentage of patients who discontinued the study during the tape treatment phase due to lack of efficacy.
Time Frame: Days 1 through Day 7 of tape treatment phase
Population: Reported data are based on Intent-to-Treat patient population.
Measure: Number; unit: percentage of patients who discontinued
Arm/Group | Placebo Tape, Daily for 12 Hours | Flurbiprofen Tape, Daily for 12 Hours | Placebo Tape, Daily for 24 Hours | Flurbiprofen Tape, Daily for 24 Hours
Number analyzed (Participants) | 20 | 42 | 22 | 43
percentage of patients who discontinued | 0 | 2.4 | 0 | 2.3

10. Secondary Outcome: Patient Assessment of Wearability of Therapy
Description: At Day 7, patients assessed the wearability of their treatment tape (ease of application, stays in place, comfortable to wear) using a 4-point scale, where:
  1 = Excellent, 4 = Poor.
Time Frame: Day 7
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Placebo Tape, Daily for 12 Hours | Flurbiprofen Tape, Daily for 12 Hours | Placebo Tape, Daily for 24 Hours | Flurbiprofen Tape, Daily for 24 Hours
Number analyzed (Participants) | 19 | 41 | 22 | 42
participants
  Ease of application, 1: Excellent | 1 | 1 | 0 | 3
  Ease of application, 2: Good | 5 | 9 | 3 | 9
  Ease of application, 3: Fair | 5 | 11 | 9 | 12
  Ease of application, 4: Poor | 8 | 20 | 10 | 18
  Stays in place, 1: Excellent | 8 | 16 | 6 | 10
  Stays in place, 2: Good | 3 | 11 | 5 | 20
  Stays in place, 3: Fair | 5 | 11 | 7 | 2
  Stays in place, 4: Poor | 3 | 3 | 4 | 10
  Comfortable to wear, 1: Excellent | 8 | 18 | 9 | 22
  Comfortable to wear, 2: Good | 8 | 14 | 8 | 14
  Comfortable to wear, 3: Fair | 0 | 9 | 2 | 2
  Comfortable to wear, 4: Poor | 3 | 0 | 3 | 4

ADVERSE EVENTS:
Time Frame: Adverse event data for the Tape Treatment phase (Days 1 - 7) are reported below.
Groups:
- Flurbiprofen Tape, Daily for 12 Hours: Two flurbiprofen tapes (one on each side of the spine) were applied on the lower back area once daily for 7 days. The tapes remained on for 12 hours of continuous treatment per day. Each tape included 31.5 mg flurbiprofen for a total daily dose of 63 mg.
Arm/Group | Placebo Tape, Daily for 12 Hours | Flurbiprofen Tape, Daily for 12 Hours | Placebo Tape, Daily for 24 Hours | Flurbiprofen Tape, Daily for 24 Hours
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/42 | 0/22 | 0/43
Other Adverse Events (participants affected / at risk) | 9/20 | 11/42 | 12/22 | 11/43
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Tape, Daily for 12 Hours (N=20) | Flurbiprofen Tape, Daily for 12 Hours (N=42) | Placebo Tape, Daily for 24 Hours (N=22) | Flurbiprofen Tape, Daily for 24 Hours (N=43)
Stomach discomfort (Gastrointestinal disorders) | 0 | 1 | 2 | 0
Application site erythema (General disorders) | 0 | 1 | 4 | 5
Application site irritation (General disorders) | 2 | 4 | 1 | 2
Application site paraesthesia (General disorders) | 1 | 0 | 0 | 0
Application site pruritus (General disorders) | 1 | 4 | 5 | 2
Application site rash (General disorders) | 2 | 1 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 2 | 1
Headache (Nervous system disorders) | 2 | 2 | 2 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
An Institution Publication may be published provided that it does not disclose Confidential Information other than the study results from Institution's study data. The proposed Institution Publication shall be submitted to sponsor for review and comment at least 30 days prior to submitting it to a third party. If sponsor requests a delay in order to file patent applications, the Institution Publication may be delayed for submission to a third party for up to 120 days after sponsor request.